# INFORMED CONSENT FORM

Determining the Effectiveness of the Geriatric Pain Measure in Older Adults Attending a Gynecology Clinic

**Document date:** 05/11/2015

NTC Number: No



# BURSA YÜKSEK İHTİSAS TRAINING AND RESEARCH HOSPITAL

## INFORMED CONSENT FORM (FOR SURVEY RESEARCH)

owment Code: EY. FR. 17

Release Date:23.11.2013 Revision Date:05.11.2015

Revision Number: 02 | Page Number: 1/2

Version Number:

### PLEASE TAKE TIME TO READ THIS DOCUMENT CAREFULLY

We invite you to a survey based on a questionnaire titled "Determination of the effectiveness of the Geriatric Pain Scale in elderly individuals who come to the gynaecology outpatient clinic" conducted by Nursel VATANSEVER, Akif BULUT and Hatice AYDIN. Before deciding whether or not to participate in this research, you need to know why and how the research will be conducted, and the potential benefits and inconveniences this research will bring to the volunteer participants. For this reason, it is very important to read and understand this form. Take time to carefully read the information below. If you want, discuss this information with your family and / or relatives. If there are things you do not understand and are not clear to you, or if you want more information, ask us. If you agree to participate in this survey, you will be given a copy of this form filled in by you and the principal investigator for you to keep.

Participation in the research is entirely voluntary. Do not be under the pressure or suggestion of anyone while answering the questions on the questionnaires provided to you. The information obtained from these forms will be used purely for research purposes and your identity information will be kept strictly confidential.

You have the right not to participate in the study or to guit at any time. In either case, there will be absolutely no penalty or loss of benefits you are entitled to.

> Research Supervisor (Name, Surname-Title-Signature)

Aim of the Study: To evaluate the effectiveness of the Geriatric Pain Scale, which is a multidimensional pain assessment method for the elderly, in elderly individuals who come to the gynaecology outpatient clinic.

Methods to be Followed and Procedures to be Followed: Within the scope of the study, Patient Information Form, Mini Mental Status Assessment Test and Geriatric Pain Scale will be collected by the researcher in the form of questions and answers on a voluntary basis.

**Duration of the Research:** 

**Expected Number of Volunteers: 100** 

Possible Benefits and Discomfort it May Bring to You: It will benefit you as an individual in the correct assessment of pain. During the execution of our study, there will be no risk or discomfort.

Research Place(s): Bursa Yüksek İhtisas Training and Research Hospital

Researchers Participating in the Research:

# BURSA YÜKSEK İHTİSAS TRAINING AND RESEARCH HOSPITAL

## INFORMED CONSENT FORM (FOR SURVEY RESEARCH)

pocument Code: EY. FR. 17

Release Date:23.11.2013 Revision Date:05.11.2015

Revision Number: 02 | Page Number: 2/2

Version Number:

### Participating in and Exiting:

Participation in this survey study is completely voluntary. You have the right not to participate in the study or to quit at any time. In addition, the responsible investigator can exclude you from the study if necessary. There will be no penalty or loss of benefits you are entitled to for not participating, leaving, or dismissed from the study.

Costs: There are no expenses in the survey process.

### Confidentiality:

The information obtained from this study will be used purely for research purposes and your identity information will be kept strictly confidential.

1,....,[name and surname of the volunteer (in their own handwriting)] read the text above and fully understood the purpose of the survey study I was asked to participate in, and my voluntary responsibilities. I had the opportunity to ask questions and discuss the survey and got satisfactory answers. I understood that I could guit this study at any time and without giving any reason, and that I would not encounter any negativity when I quit.

Under these circumstances, I agree to participate in the survey study in question (I agree to my child/guardian's participating in this study) without any pressure or coercion.

| Volunteer's (In his/her own handwriting) Name-Surname: |
|--------------------------------------------------------|
| Signature: |
| Address: (Telephone No, Fax No, if available): |
| Date (day / month / year):/ |

For Those Under Guardianship or Custody Parent or Guardian's (in his own handwriting) Name-Surname:

Signature:

Address:

(Telephone No, Fax No, if available):

Date (day / month / year): ..../..../

The Researcher Making the Statements

Name-Surname:

Signature:

Date (day / month / year): ..../..../

The Institution Officer Witnessing the Approval Process from the Beginning to the End (Studies in the clinic are valid for survey studies)

Name-Surname:

Signature:

Dutv:

Date (day / month / year): ..../..../